CLINICAL TRIAL: NCT07175285
Title: Prospective, Observational Study in Participants With Active Systemic Lupus Erythematosus (SLE) (Including Lupus Nephritis) With Inadequate Response to Glucocorticoids and At Least 2 Immunosuppressants
Brief Title: A Study in Participants With Active Systemic Lupus Erythematosus With Inadequate Response to Glucocorticoids and ≥2 Immunosuppressants
Acronym: BENCHMARK-SLE
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA061-1025
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Systemic lupus erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Participants with systemic lupus erythematosus (SLE), including Lupus Nephritis, with inadequate response to glucocorticoids and at least 2 immunosuppressants, receiving current standard of care treatment options.
  Interventions: Drug: Current standard of care treatment options

INTERVENTIONS:
Drug: Current standard of care treatment options — According to the product label

SUMMARY:
The purpose of this study is to characterize the efficacy and safety of current standard of care treatment options in participants with active systemic lupus erythematosus (SLE; including lupus nephritis) with inadequate response to glucocorticoids and at least two immunosuppressants

ELIGIBILITY:
Inclusion Criteria:

* Participants must have signed and dated an Institutional Review Board/ Independent Ethics Committee (IRB/IEC)-approved written informed consent form (ICF) in accordance with regulatory, local, and institutional guidelines
* Participants must be ≥16 years of age at the time of signing the ICF
* Meet the European League Against Rheumatism (EULAR) / American College of Rheumatology (ACR) 2019 classification criteria for systemic lupus erythematosus (SLE)
* Have an inadequate response to glucocorticoids and ≥ 2 immunosuppressant therapies such as cyclophosphamide, mycophenolic acid and its derivatives, belimumab, anifrolumab, rituximab, methotrexate, azathioprine, obinutuzumab, cyclosporine, tacrolimus, or voclosporin, used for at least 3 months each. Eligibility is regardless of prior hydroxychloroquine or any anti-malarial treatment. Inadequate response is defined as a lack of response, insufficient response, or lack of sustained response after at least 3-month treatment with appropriate doses of a standard of care agent. Intolerance or contraindication may be considered as inadequate response provided it is documented and confirmed acceptable by the Adjudication Committee
* Have active disease at study entry when signing ICF, defined as:

  * ≥ 1 British Isles Lupus Assessment Group Index (BILAG) A OR ≥ 1 BILAG B with history of SLE manifestations that would qualify for a BILAG A within the last 24 months, AND
  * Positive autoantibodies (at least one) to confirm diagnosis of SLE: Antinuclear antibody ≥1:160, anti-dsDNA, anti-Sm, anti-Ro (SSA), anti-La (SSB), or low complement (C3 or C4)
* Participants with lupus nephritis meeting the study eligibility criteria must have had a renal biopsy per standard of care within the last 6 months indicating the presence of active Class III or IV lupus glomerulonephritis (alone or in combination with Class V) according to the 2018 Revised International Society of Nephrology/Renal Pathology Society (ISN/RPS), with < 60% interstitial fibrosis and tubular atrophy < 60% global glomerulosclerosis

Exclusion Criteria:

* Pregnant women
* Participants enrolled in concurrent interventional clinical trials involving investigational therapies or any other clinical trial
* Participant is unwilling and unable to adhere to the study visit schedule and other protocol requirements

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include individuals diagnosed with systemic lupus erythematosus (SLE) with inadequate response (a lack of response, insufficient response, or lack of sustained response after at least 3-month treatment with appropriate doses of a standard of care therapy) to glucocorticoids and at least two immunosuppressants according to routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 223 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2032-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of of participants achieving Definition of Remission in Systemic Lupus Erythematosus (DORIS) at 6 months along with the 95% CI. | 6 months

SECONDARY OUTCOMES:
Number of participants achieving drug-free Definition of Remission in Systemic Lupus Erythematosus (DORIS) remission | At 12, 24, 36, 48, and 60 months
Complete renal response (CRR) for participants with baseline lupus nephritis (LN) | At 6, 12, 24, 36, 48, and 60 months
Lupus-Low Disease Activity State (LLDAS) for participants with baseline Systemic Lupus Erythematosus Disease Activity Questionnaire (SLEDAI) ≥ 6 | At 12, 24, 36, 48, and 60 months
Incidence and severity of flares, as assessed by Systemic Lupus Erythematosus Disease Activity Questionnaire (SLEDAI) index | Up to 60 months
SLE Responder Index 4 (SRI-4) for participants with baseline Lupus Erythematosus Disease Activity Questionnaire (SLEDAI) ≥ 6 | At 6, 12, 24, 36, 48, and 60 months
Change from baseline in proteinuria and estimated glomerular filtration rate (eGFR) - of those with high proteinuria and low eGFR | At 6, 12, 24, 36, 48, and 60 months
Change in 2012 Systemic Lupus Collaborating Clinics Criteria for SLE (SLICC) damage from baseline | At 12, 24, 36, 48, and 60 months
Number of participants that maintain remission status as assessed by DORIS, LLDAS, and SRI-4 | At 6, 12, 24, 36, 48, and 60 months
  Definition of Remission in Systemic Lupus Erythematosus (DORIS), Lupus-Low Disease Activity State (LLDAS) and SLE Responder Index 4 (SRI-4)
Duration of treatment response | Up to 60 months
Time to treatment response | Up to 60 months
Incidence of adverse events (AEs) including serious AEs | Up to 60 months
Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) patient reported outcome (PRO) from baseline | Baseline, and at 6, 12, 24, 36, 48, and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (41):
- United States (17):
  - Local Institution - 0062, Mesa, Arizona
  - Local Institution - 0054, La Jolla, California
  - Rheumatology Center of San Diego, San Diego, California
  - Local Institution - 0063, Fort Lauderdale, Florida
  - Local Institution - 0061, Hollywood, Florida
  - LIFE Clinical Trials, Margate, Florida
  - Local Institution - 0064, Rockville, Maryland
  - Local Institution - 0034, Ann Arbor, Michigan
  - AA MRC, Grand Blanc, Michigan
  - Local Institution - 0060, West Long Branch, New Jersey
  - Local Institution - 0039, Brooklyn, New York
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Local Institution - 0037, Durham, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Local Institution - 0052, Philadelphia, Pennsylvania
  - El Paso Medical Research Institute (MedResearch, Inc), El Paso, Texas
  - Local Institution - 0051, Van Vleck, Texas
- Argentina (2):
  - Local Institution - 0029, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0050, Buenos Aires
- Local Institution - 0042, São Paulo, Brazil
- Canada (2):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Local Institution - 0038, Sherbrooke, Quebec
- France (2):
  - Local Institution - 0023, Bordeaux
  - Local Institution - 0044, Paris
- Germany (2):
  - Local Institution - 0041, Kiel, Schleswig-Holstein
  - Local Institution - 0043, Mainz
- Israel (2):
  - Meir Medical Center, Kfar Saba, M
  - Carmel Medical Center, Haifa
- Italy (2):
  - Local Institution - 0040, Ferrara, RE
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino, TO
- Japan (3):
  - Local Institution - 0049, Kitakyushu-shi, Fukuoka
  - Local Institution - 0053, Sendai, Miyagi
  - Local Institution - 0055, Wakayama
- Local Institution - 0046, San Juan, PR, Puerto Rico
- Spain (2):
  - Local Institution - 0047, Mérida, Badajoz
  - Local Institution - 0048, Barcelona
- United Kingdom (5):
  - Local Institution - 0056, Oxford, OXF
  - Local Institution - 0058, Bath, SOM
  - Local Institution - 0045, Wolverhampton, West Midlands
  - Local Institution - 0059, London
  - Local Institution - 0057, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts